CLINICAL TRIAL: NCT01356823
Title: A Randomized, Double-Blinded, Placebo-Controlled, Dose-Ranging Study of Recombinant Human Papillomavirus Virus 16/18 Bivalent Vaccine (E.Coli)in Healthy Female Subjects Aged 18 to 25 Years
Brief Title: Dose-Ranging Study of Recombinant Human Papillomavirus Virus 16/18 Bivalent Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xiamen University (Other)
Collaborators: Xiamen Innovax Biotech Co., Ltd (Industry); Beijing Wantai Biological Pharmacy Enterprise Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jun Zhang, professor, Xiamen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HPV-PRO-002
Record Dates: First submitted 2011-05-13; First posted 2011-05-20 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2014-02

CONDITIONS: Cervical Intraepithelial Neoplasia; Cervical Cancer
Keywords: Human Papilloma Virus 16; Human Papilloma Virus 18; vaccine; Cervical Intraepithelial Neoplasia; cervical Cancer
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms | interventions — Papillomavirus Vaccines; Hepatitis B Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 30μg HPV (Experimental): Participants in this arm would receive 30μg HPV vaccines which contains 20μg HPV 16 antigen and 10μg HPV 18 antigen
  Interventions: Biological: 30μg HPV
- 60μg HPV (Experimental): Participants in this arm would receive 60μg HPV vaccines which contains 40μg HPV 16 antigen and 20μg HPV 18 antigen
  Interventions: Biological: 60μg HPV
- 90μg HPV (Experimental): Participants in this arm would receive 90μg HPV vaccines which contains 60μg HPV 16 antigen and 30μg HPV 18 antigen
  Interventions: Biological: 90μg HPV
- hepatitis B vaccine (Placebo Comparator): Participants in this arm would receive hepatitis B vaccine.
  Interventions: Biological: Hepatitis B vaccine

INTERVENTIONS:
Biological: 30μg HPV — Participants would intramuscularly receive 30μg of HPV 16/18 bivalent vaccine at 0, 1, 6 month for 3 doses.
  Arms: 30μg HPV
Biological: 60μg HPV — Participants would intramuscularly receive 60μg of HPV 16/18 bivalent vaccine at 0, 1, 6 month for 3 doses.
  Arms: 60μg HPV
Biological: 90μg HPV — Participants would receive 90μg HPV vaccines which contains 60μg HPV 16 antigen and 30μg HPV 18 antigen
  Arms: 90μg HPV
Biological: Hepatitis B vaccine — Participants would intramuscularly receive 10μg of hepatitis B vaccine at 0, 1, 6 month for 3 doses.
  Arms: hepatitis B vaccine

SUMMARY:
This is a phase II clinical study of the novel recombinant HPV 16/18 bivalent vaccine expressed in E. coli.

The primary purpose of this study is to evaluate which dosage of the HPV vaccine can induce higher antibody and at the same time caused less adverse events.

The secondary purpose of this study is to to evaluate the safety and immunopersistence of the study vaccine.

DETAILED DESCRIPTION:
Totally 1600 healthy women of 18-25 years of age were enrolled. The participants were randomly stratified into 4 groups and receive different dosage of human papillomavirus (HPV) vaccine or placebo administered intramuscularly according to a 0-1-6 month schedule. The women were actively monitored for adverse events for 1 month after each injection. Severe adverse events during the trial were followed up. Serum samples from all the subjects would be collected on day 0, 7m, 24m, 48m and 72m to evaluate the immunogenicity and immuno-persistency.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from the subject prior to enrolment;
* Female between, and including, 18 and 25 years of age at the time of enrolment;
* Subjects must be free of obvious health problems;
* Not pregnant and having no plan for pregnancy;

Exclusion Criteria:

* Pregnant or breastfeeding or having plan for pregnancy during the whole study (Month 0-7);
* Previous vaccination against HPV;
* Having severe allergic history or other immunodeficiency;
* Chemotherapy and other immunosuppressive agents using;

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1600 (Actual)
Dates: Start 2011-03; Primary Completion 2011-12 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Seroconversion of anti-HPV 16 and anti-HPV 18 neutralizing antibody | 7 months
  To detect the anti-HPV 16 and anti-HPV 18 neutralizing antibody level on day 1 and one month after dose 3.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | 7 months
  All the adverse events in one month after each dose would be recorded in the diary card. All the Serious Adverse Events(SAE) occurred during clinical trial time frame would be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, Master, Study Chair — Xiamen University; Yuemei Hu, Bachelor, Principal Investigator — Jiangsu Provincial Centre for Disease Control and Prevention; Ting Wu, Ph. D, Study Director — Xiamen University
Locations (1):
- Jiangsu Provincial Centre for Disease Control and Prevention, Nanjing, Jiangsu, China

REFERENCES:
- [Result] Wu T, Hu YM, Li J, Chu K, Huang SJ, Zhao H, Wang ZZ, Yang CL, Jiang HM, Wang YJ, Lin ZJ, Pan HR, Sheng W, Wei FX, Li SW, Wang Y, Zhu FC, Li CG, Zhang J, Xia NS. Immunogenicity and safety of an E. coli-produced bivalent human papillomavirus (type 16 and 18) vaccine: A randomized controlled phase 2 clinical trial. Vaccine. 2015 Jul 31;33(32):3940-6. doi: 10.1016/j.vaccine.2015.06.052. Epub 2015 Jun 19. PMID 26100924